CLINICAL TRIAL: NCT05465837
Title: Comparison Between Early and Late Tracheostomy in ICU Patients Including Non-Covid and Covid Patients, an Observational Cohort Study at SQUH
Brief Title: Comparison Between Early and Late Tracheostomy in Non-Covid and Covid
Acronym: CELT
Status: Completed | Type: Observational
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Other Study IDs: MREC#2688
Record Dates: First submitted 2022-07-03; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: Non-Covid; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non covid Tracheostomy Patients: Adult patients (>18 years) who underwent tracheostomy without having the covid-19 infection
  Interventions: Procedure: Tracheostomy
- Covid-19 Tracheostomy Patients: Adult patients (>18 years) who underwent tracheostomy had the covid-19 infection
  Interventions: Procedure: Tracheostomy

INTERVENTIONS:
Procedure: Tracheostomy — Early and Late Tracheostomy (</= 10 days: Early and >10 days: Late)

SUMMARY:
Tracheostomy is commonly indicated for the patient who is requiring long period of mechanical ventilation. Patient who require mechanical ventilation for >10 days and longer mostly get tracheostomized. Tracheostomy is associated with less complications associated with endotracheal intubation. Tracheostomy is a surgical procedure whereby an external artificial opening is made in the trachea. Several techniques are used to perform tracheostomy, including the classical standard surgical procedure completed in a surgical room and the percutaneous method performed at the patient's bedside. Surgical and percutaneous procedures are usually performed by different surgical specialists such as general; thoracic; ear, nose and throat (ENT); or maxillofacial surgeons, but percutaneous procedures are usually but not exclusively performed by surgeons and intensivists.

Early tracheostomy might reduce the length of ICU stay, whereas delaying the tracheostomy might avoid a few. A review of recent studies showed a decrease in the mortality rate in early tracheostomised patients compared with late. Tracheostomy is a routine bedside procedure in ICU with minimal complications.

Severe acute respiratory syndrome (SARS) and Coronavirus 2 (SARS-CoV-2) started to appear in Oman in early February 2020, resulting in an escalation of new cases within days. In the first weeks of the pandemic, many guidelines from different specialties recommended avoiding early tracheostomy to minimize the risk of infection to clinicians.

Specifically, recommendations for tracheostomy in the current pandemic were rooted in the assumption that maximal infectivity of this novel virus occurred around day 7 to 10 after symptom onset, and performing tracheostomy at that time would endanger maximal risk to those performing it. Hence these factors interfered with the timing of Tracheostomy for Covid patients.

This is an observational cohort study. It will assess patients admitted to ICU at SQUH during the period between January 2020 and December 2021 with Non-Covid and Covid-19 patients. This study will assess the causes and outcomes of early and late tracheostomy in Non-Covid and Covid-19 patients requiring mechanical ventilation. Main outcomes will include mortality rate, ventilation days, and ICU length of stay.

DETAILED DESCRIPTION:
Introduction:- Tracheostomy is a common procedure for critically ill patients who require long-term mechanical ventilation (3) and have a low Glasgow coma scale and for chest toileting. Compared with an endotracheal tube, a shorter tracheostomy tube that bypasses the mouth and pharynx can avoid oropharyngeal and laryngeal complications, improve patient comfort and reduce sedative drug use.

Early versus late tracheostomy:

In one study comparing early and late tracheostomy, they included eight RCTs. Results showed moderate quality from seven RCTs and lower mortality rates in the early as compared with the late tracheostomy group. On the other hand, in another study which was a prospective observational study, the results showed that there was no difference in 3-month mortality between early and late tracheostomy.

Covid-19 is a recently emerged disease and has resulted in an increasing number of patients requiring mechanical ventilation and ICU admission. Several recommendations and guidelines have discussed when to perform a tracheostomy in COVID-19 patients, while the timing is varied across the literature. Recommendations from the UK and North America suggested that tracheostomy should be delayed until at least 14 days from endotracheal intubation to clarify prognostic information and for the viral load to sufficiently decline. On the other hand, early tracheostomy may help in early weaning (around 7-10 days))

In this study, we aimed to investigate the differences in outcomes when tracheostomy is done early versus late in covid and non-covid cases.

Aim of the Study:

The aim of the current study is to analyze the outcomes of patients with confirmed SARS-CoV-2 pneumonia who underwent tracheostomies and explore the association between the timing of tracheostomy and the outcomes of these patients and compare them with Non-Covid-19 patients.

. The primary outcomes: Mortality in Covid versus Non-Covid cases The secondary outcomes: Ventilation days and ICU length of stay in Covid versus Non-Covid cases.

Methodology:- This retrospective study will be conducted in Sultan Qaboos University Hospital, Oman. After taking Ethics approval, all patients who undergo tracheostomy in intensive care units (ICUs) at SQUH from January 1, 2020, to December 2021 will be screened. A list of all patients who underwent tracheostomies during the study period will be obtained from the Hospital Information system. Their electronic patient records will be scanned, and data will be obtained.

Study Population:

Inclusions:

• Adult ICU patients (more than 18 years old) who underwent tracheostomy in ICU.

Exclusions:

• Tracheostomy performed as part of operative management.

Study Design and Methods:

Overview: This retrospective, observational cohort study will assess the outcomes of early and late tracheostomy in Non-Covid and Covid patients.

Sample size: All tracheostomized patients during the study period will be included in the study.

Study Method:

Medical records of patients will be reviewed, and data will be collected by investigators. Sociodemographic and clinical data will be collected for all patients, including age, sex, medical history, technique and day of ventilation days, ICU length of stay, and mortality.

Details of the tracheostomy procedure, including timing, type (percutaneous or surgical), and complications, will be noted.

Justification of the current study:

In this study, we intend to analyze the outcomes of early and late tracheostomy in covid and non-covid patients. We hope to find a strategy for choosing an appropriate time for tracheostomy in covid and non-covid patients, which will give better outcomes and help reduce ICU mortality, ventilator days, and length of stay.

ETHICAL Aspects:

The master chart will not carry patient names and even MRN will not be accessible to anyone except the principal investigator. In the end, the study subjects will be given code numbers in the final master chart and their ID will not be revealed to the statistician.

Data Management and Analyses:

Statistical analysis: Normally distributed and non-normally distributed continuous variables will be presented as the mean (SD) and median [IQR], respectively. Categorical variables are presented as numbers (%). Early tracheostomy will be defined as tracheostomy within 10 days of intubation, and late tracheostomy will be defined as tracheostomy after 10 days. All statistical analyses will be performed using the SPSS software system.

ELIGIBILITY:
Inclusion Criteria:

* • Adult ICU patients (more than 18 years old) who underwent tracheostomy in ICU.

Exclusion Criteria:

* • Tracheostomy performed as part of operative management.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Population > 18 years old, admitted to Non-Covid and Covid-19 ICU OF Sultan Qaboos University Hospital, Oman, who got tracheostomized during their stay in ICU
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Mortality in Covid versus Non-Covid cases | upto 90 days
  30 and 60 Days mortality

SECONDARY OUTCOMES:
Ventilation days | upto 90 days
  Number of ventilation days
ICU length of stay | upto 90 days
  ICU length of stay total

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Burad, Principal Investigator — Sultan Qaboos University Hospital
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be deposited to Repository: Mendeley and will be made available after this study is published
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be made available after this study is published (after a few months of publication, up to 5 years)
Access Criteria: Will be provided to a researcher interested and writes to the Principal investigator about the need for the data

REFERENCES:
- [Background] Givi B, Schiff BA, Chinn SB, Clayburgh D, Iyer NG, Jalisi S, Moore MG, Nathan CA, Orloff LA, O'Neill JP, Parker N, Zender C, Morris LGT, Davies L. Safety Recommendations for Evaluation and Surgery of the Head and Neck During the COVID-19 Pandemic. JAMA Otolaryngol Head Neck Surg. 2020 Jun 1;146(6):579-584. doi: 10.1001/jamaoto.2020.0780. PMID 32232423
- [Background] He X, Lau EHY, Wu P, Deng X, Wang J, Hao X, Lau YC, Wong JY, Guan Y, Tan X, Mo X, Chen Y, Liao B, Chen W, Hu F, Zhang Q, Zhong M, Wu Y, Zhao L, Zhang F, Cowling BJ, Li F, Leung GM. Temporal dynamics in viral shedding and transmissibility of COVID-19. Nat Med. 2020 May;26(5):672-675. doi: 10.1038/s41591-020-0869-5. Epub 2020 Apr 15. PMID 32296168
- [Background] Scales DC, Ferguson ND. Tracheostomy: it's time to move from art to science. Crit Care Med. 2006 Dec;34(12):3039-40. doi: 10.1097/01.CCM.0000242924.24342.9D. No abstract available. PMID 17130697
- [Background] Polok K, Fronczek J, van Heerden PV, Flaatten H, Guidet B, De Lange DW, Fjolner J, Leaver S, Beil M, Sviri S, Bruno RR, Wernly B, Artigas A, Pinto BB, Schefold JC, Studzinska D, Joannidis M, Oeyen S, Marsh B, Andersen FH, Moreno R, Cecconi M, Jung C, Szczeklik W; COVIP study group. Association between tracheostomy timing and outcomes for older critically ill COVID-19 patients: prospective observational study in European intensive care units. Br J Anaesth. 2022 Mar;128(3):482-490. doi: 10.1016/j.bja.2021.11.027. Epub 2021 Nov 29. PMID 34955167
- [Background] Bosel J, Schiller P, Hook Y, Andes M, Neumann JO, Poli S, Amiri H, Schonenberger S, Peng Z, Unterberg A, Hacke W, Steiner T. Stroke-related Early Tracheostomy versus Prolonged Orotracheal Intubation in Neurocritical Care Trial (SETPOINT): a randomized pilot trial. Stroke. 2013 Jan;44(1):21-8. doi: 10.1161/STROKEAHA.112.669895. Epub 2012 Nov 29. PMID 23204058
- [Background] Hsu CL, Chen KY, Chang CH, Jerng JS, Yu CJ, Yang PC. Timing of tracheostomy as a determinant of weaning success in critically ill patients: a retrospective study. Crit Care. 2005 Feb;9(1):R46-52. doi: 10.1186/cc3018. Epub 2004 Dec 23. PMID 15693966
- [Result] Andriolo BN, Andriolo RB, Saconato H, Atallah AN, Valente O. Early versus late tracheostomy for critically ill patients. Cochrane Database Syst Rev. 2015 Jan 12;1(1):CD007271. doi: 10.1002/14651858.CD007271.pub3. PMID 25581416